CLINICAL TRIAL: NCT01908231
Title: Prognostic Value of Plasma Lactate Levels Among Patients With Acute Pulmonary Embolism: the Thrombo-Embolism Lactate Outcome Study
Brief Title: Prognostic Value of Plasma Lactate Levels Among Patients With Acute Pulmonary Embolism
Acronym: TELOS
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Simone Vanni, MD, PhD, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 0313
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism, plasma lactate, right ventricular dysfunction
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary Embolism: Consecutive adult patients (minimum age eighteen) who presented to the ED of the hospitals participating in the study with clinical suspicion of PE will be considered for the study. We excluded patients with life expectancies of less than 3 months, and patients with first symptoms 15 days or more before inclusion.

SUMMARY:
To prospectively investigate the association between plasma lactate concentration and short-term adverse outcomes in patients with acute PE.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) represents 0.4% of hospitalizations and is the third leading cause of death due to cardiovascular disease (1). In contrast to stroke and acute coronary syndromes, its mortality has not decreased in recent decades likely due to only minor advances in short-term prognostication and treatment strategies (2).The presence of shock or hypotension remains the principal prognostic clinical marker and,to date, is the only factor that clearly indicates a more aggressive treatment than heparin (3). However, only 5% of patients with acute PE present with shock. The majority of PE patients are normotensive and are usually treated with heparin alone. Several studies have looked for new prognostic indicators in order to better stratify normotensive PE patients. A large body of evidence shows that right ventricular dysfunction/injury markers such as elevation of brain natriuretic peptides, troponins, and echocardiographic evidence of right ventricular dysfunction (RVD) are associated with adverse prognosis (3-8). However, these markers have some important limitations. Echocardiography is usually not available around-the-clock in most clinical settings, moreover it shares with troponins and natriuretic peptides a good negative predictive value (>90%) but a low positive predictive value (about 10%) for short-term mortality, probably precluding these markers' usefulness to target more aggressive treatments (8).

Plasma lactate concentration is a marker of the severity of the tissue oxygen supply-to-demand imbalance. It may reflect tissue hypoperfusion also in the presence of normal blood pressure. Accordingly, in other critical settings such as sepsis,plasma lactate concentration is considered to be an accurate prognostic marker as it rises before hemodynamic impairment is clinically evident (9). Furthermore, plasma lactate concentration can be easily and rapidly assayed on arterial blood samples using a blood gas analyzer, which is usually available in emergency departments (EDs) and intensive care units. Recently, a retrospective study showed that plasma lactate ≥ 2 mmol/L was associated with a high mortality rate in patients with acute PE (10). Moreover a prospective monocentric study confirmed these retrospective results and revealed that plasma lactate has prognostic relevance beyond known clinical and instrumental prognostic markers (TELOS study, Ann Emerg Med, in press, see attached file)

The aim of present study is to prospectively investigate the association between plasma lactate concentration and short-term adverse outcomes in patients with acute PE. In particular, we examine whether high plasma lactate (≥ 2 mmol/L) is associated with a high incidence of PE related major adverse events, defined as PE related death or hemodynamic collapse >10% within 7 days of follow-up. Moreover we investigate whether plasma lactate shows incremental prognostic value to clinically overt hemodynamic impairment and to RVD/injury markers, maintaining prognostic relevance in both hypotensive and normotensive PE patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic objective pulmonary embolism

Exclusion Criteria:

* life expectancies of less than 3 months
* first symptoms 15 day or more before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (minimum age eighteen) who presented to the ED of the hospitals participating in the study with clinical suspicion of PE will be considered for the study. We excluded patients with life expectancies of less than 3 months, and patients with first symptoms 15 day or more before inclusion.
  The diagnosis of PE will be established by spiral computed tomography or by lung scan or a selective pulmonary angiogram.
  Patients with proven PE who will give written consent to the use of their medical information for research purposes will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The composite of PE related death or hemodynamic collapse | 7 days.
  PE related death was defined as a fatal event occurring in the hours after clinical deterioration due to PE, including an objectively diagnosed recurrent PE, or if death could not be attributed to a documented cause and PE could not be confidently ruled out. Autopsy is not mandatory.
  Hemodynamic collapse is defined as at least 1 of the following: (i) the need for cardiopulmonary resuscitation; (ii) systolic blood pressure <90 mm Hg for at least 15 minutes, or drop of systolic blood pressure by at least 40 mm Hg for at least 15 minutes, with signs of end-organ hypoperfusion (cold extremities, or urinary output <30 mL/h, or mental confusion); (iii) the need for catecholamines (except for dopamine at a rate of < 5 μg kg-1 min-1) to maintain adequate organ perfusion and a systolic blood pressure of >90 mm Hg; (iiii) the need for invasive or noninvasive mechanical ventilation; (iiiii) imaging-confirmed symptomatic recurrence of PE within 7 days.

SECONDARY OUTCOMES:
all cause death | 30 days
PE recurrence | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Grifoni, MD, Study Chair — Emergency department, Azienda Ospedaliero Universitaria Careggi
Locations (4):
- Italy (3):
  - Azienda Ospedaliero Universitaria Careggi, Emergency Department, Florence
  - Presidio Ospedaliero Livorno, Livorno
  - Azienda ospedaliera universitaria San Giovanni Battista (Molinette), Torino
- Respiratory Department and Medicine Department, Ramón y Cajal Hospital and Alcalá de Henares University, Madrid, Spain

REFERENCES:
- [Background] Pulido T, Aranda A, Zevallos MA, Bautista E, Martinez-Guerra ML, Santos LE, Sandoval J. Pulmonary embolism as a cause of death in patients with heart disease: an autopsy study. Chest. 2006 May;129(5):1282-7. doi: 10.1378/chest.129.5.1282. PMID 16685020
- [Background] Burge AJ, Freeman KD, Klapper PJ, Haramati LB. Increased diagnosis of pulmonary embolism without a corresponding decline in mortality during the CT era. Clin Radiol. 2008 Apr;63(4):381-6. doi: 10.1016/j.crad.2007.10.004. Epub 2007 Dec 21. PMID 18325357
- [Background] Torbicki A, Perrier A, Konstantinides S, Agnelli G, Galie N, Pruszczyk P, Bengel F, Brady AJ, Ferreira D, Janssens U, Klepetko W, Mayer E, Remy-Jardin M, Bassand JP; ESC Committee for Practice Guidelines (CPG). Guidelines on the diagnosis and management of acute pulmonary embolism: the Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). Eur Heart J. 2008 Sep;29(18):2276-315. doi: 10.1093/eurheartj/ehn310. Epub 2008 Aug 30. PMID 18757870
- [Background] Grifoni S, Olivotto I, Cecchini P, Pieralli F, Camaiti A, Santoro G, Conti A, Agnelli G, Berni G. Short-term clinical outcome of patients with acute pulmonary embolism, normal blood pressure, and echocardiographic right ventricular dysfunction. Circulation. 2000 Jun 20;101(24):2817-22. doi: 10.1161/01.cir.101.24.2817. PMID 10859287
- [Background] Kucher N, Goldhaber SZ. Cardiac biomarkers for risk stratification of patients with acute pulmonary embolism. Circulation. 2003 Nov 4;108(18):2191-4. doi: 10.1161/01.CIR.0000100687.99687.CE. No abstract available. PMID 14597581
- [Background] Kline JA, Zeitouni R, Marchick MR, Hernandez-Nino J, Rose GA. Comparison of 8 biomarkers for prediction of right ventricular hypokinesis 6 months after submassive pulmonary embolism. Am Heart J. 2008 Aug;156(2):308-14. doi: 10.1016/j.ahj.2008.03.026. Epub 2008 Jun 18. PMID 18657661
- [Background] Binder L, Pieske B, Olschewski M, Geibel A, Klostermann B, Reiner C, Konstantinides S. N-terminal pro-brain natriuretic peptide or troponin testing followed by echocardiography for risk stratification of acute pulmonary embolism. Circulation. 2005 Sep 13;112(11):1573-9. doi: 10.1161/CIRCULATIONAHA.105.552216. Epub 2005 Sep 6. PMID 16144990
- [Background] Shapiro NI, Trzeciak S, Hollander JE, Birkhahn R, Otero R, Osborn TM, Moretti E, Nguyen HB, Gunnerson KJ, Milzman D, Gaieski DF, Goyal M, Cairns CB, Ngo L, Rivers EP. A prospective, multicenter derivation of a biomarker panel to assess risk of organ dysfunction, shock, and death in emergency department patients with suspected sepsis. Crit Care Med. 2009 Jan;37(1):96-104. doi: 10.1097/CCM.0b013e318192fd9d. PMID 19050610
- [Background] Vanni S, Socci F, Pepe G, Nazerian P, Viviani G, Baioni M, Conti A, Grifoni S. High plasma lactate levels are associated with increased risk of in-hospital mortality in patients with pulmonary embolism. Acad Emerg Med. 2011 Aug;18(8):830-5. doi: 10.1111/j.1553-2712.2011.01128.x. PMID 21843218
- [Background] Vanni S, Polidori G, Vergara R, Pepe G, Nazerian P, Moroni F, Garbelli E, Daviddi F, Grifoni S. Prognostic value of ECG among patients with acute pulmonary embolism and normal blood pressure. Am J Med. 2009 Mar;122(3):257-64. doi: 10.1016/j.amjmed.2008.08.031. PMID 19272487
- [Background] Grifoni S, Vanni S, Magazzini S, Olivotto I, Conti A, Zanobetti M, Polidori G, Pieralli F, Peiman N, Becattini C, Agnelli G. Association of persistent right ventricular dysfunction at hospital discharge after acute pulmonary embolism with recurrent thromboembolic events. Arch Intern Med. 2006 Oct 23;166(19):2151-6. doi: 10.1001/archinte.166.19.2151. PMID 17060547